CLINICAL TRIAL: NCT01703130
Title: Determining the Minimal Effective Volume (MEAV95) for Interscalene Brachial Plexus Block for Surgical Anesthesia
Acronym: MEAV 95
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Dr. Colin McCartney, Staff Anesthesiologist and Director of Research, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 126-2012
Record Dates: First submitted 2012-10-04; First posted 2012-10-10 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Shoulder Pain
Keywords: ISPB; Brachial Plexus Block; Anesthesia; Pain Management; Surgery
MeSH Terms: conditions — Shoulder Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Local Anesthestic Dose (Experimental)
  Interventions: Procedure: Dose of of ropivacaine 0.75% used in block procedure

INTERVENTIONS:
Procedure: Dose of of ropivacaine 0.75% used in block procedure

SUMMARY:
Interscalene block (ISB) consistently demonstrates superior pain relief after shoulder surgery. However, patients can experience complications such as blurred vision, hoarseness and shortness of breath with the standard volumes of local anesthetic used in contemporary practice. Patients with respiratory diseases are precluded because of the potential effects on respiration. However, they are then exposed to the risks of general anesthesia and opioid medications which can also have detrimental effects on respiration. Ultrasound guided ISB can reduce the local anesthetic volume required to produce anesthesia for shoulder surgery; this may reduce the complications from ISB to allow patients previously unable to benefit to have this technique, such as patients with obesity and respiratory disease. In order to do so the investigators will use an up-down methodology to find the minimum volume of local anesthetic to provide sufficient anesthesia for shoulder surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective arthroscopic shoulder surgery in the sitting position
* Patients aged >=18 and <=75 years
* ASA I-III

Exclusion Criteria:

* Patient refusal for surgery under ISBPB with sedation
* Lack of capacity to provide informed consent
* Pre-existing COPD, unstable asthma or diaphragmatic dysfunction
* Coagulopathy
* Infection at injection site
* Allergy to local anesthetics
* Opioid tolerance (>30mg oral morphine or equivalent/day for >1 week)
* BMI>40
* Inability to complete questionnaires and assessments (consent, follow-up phone call) due to language barrier
* Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
MEAV95 of ropivacaine 0.75% | 30 minutes post injection
  to determine the MEAV95 of ropivacaine 0.75% at the level of root C5-6 using the dose-finding protocol. The success of surgical anesthesia is defined by the presence of sensory blockade (no sensation/score of 0 to pinprick testing) 30 minutes post injection of local anesthetic

SECONDARY OUTCOMES:
Motor blockade | 30 minutes
  The C5 myotome covers the deltoid muscle (the most powerful motion being shoulder abduction) and the biceps brachii muscle. Biceps brachii is also innervated by C6. Therefore, motor blockade will be assessed by testing shoulder abduction and forearm flexion. Motor function will be classified as present (any movement) or absent (no movement)
Bedside spirometry | 30 minutes post block, 30min post-surgery, and 2 hours post surgery
  Bedside spirometry (FEV1, FVC, PEFR) and Pulse oximetry on air: at baseline, 30 minutes post block, 30min post-surgery, and 2 hours post surgery
Diaphragmatic excursion | 30 minutes post block, and 2 hours post surgery
  Diaphragmatic excursion: ultrasound examination at baseline, 30 minutes post block, and 2 hours post surgery
Complications | 30 minutes
  Complications: Hoarseness, Horner's syndrome, intravascular injection
Pain Scores on Visual Analog Scale | at baseline, after surgery at 30 and 60 minutes in the PACU, and at 1 hour intervals until discharge
  Visual analog scale (VAS) - at baseline, after surgery at 30 and 60 minutes in the PACU, and at 1 hour intervals until discharge
Total opioid consumption until discharge | 24 hours (at discharge)
  Total opioid consumption until discharge
Opioid related side effects | 24 hours (at discharge)
  Opioid related side effects: nausea, vomiting, dizziness, pruritis
Time to first analgesic use | within 24 hours post surgery
  Time to first analgesic use in hospital and after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Colin McCartney, Principal Investigator — Sunnybrook Health Sciences Centre; Stephen Choi, Study Chair — Sunnybrook Health Sciences Centre; Jane Wang, Study Chair — Sunnybrook Health Sciences Centre; Moein Tavakkoli Zadeh, Study Chair — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre - Holland Orthopaedic and Arthritic Centre, Toronto, Ontario, Canada

REFERENCES:
- See also: Facility website — http://sunnybrook.ca/research/